CLINICAL TRIAL: NCT06259370
Title: Benefits of Wearable Acceleration-Monitored Simulated Vigorous Intermittent Lifestyle Physical Activity (VILPA) in Young Adults
Brief Title: Benefits of VILPA in Young Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xiao-dong Zhuang (Other)
Responsible Party: Sponsor-Investigator, Xiao-dong Zhuang, Clinical Professor, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: K001
Record Dates: First submitted 2024-01-19; First posted 2024-02-14 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Activity, Motor; Health Behavior
Keywords: vigorous intermittent lifestyle physical activity; wearable device; Isokinetic strength testing
MeSH Terms: conditions — Motor Activity; Health Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- intervention group (Experimental): The intervention measures encompass the implementation of simulated vigorous intermittent lifestyle physical activity for all participants. The specific exercise regimen involves performing rope jumping activities three times a day, with each session aimed at surpassing the exercise threshold (not conducted in a continuous manner), where the heart rate should exceed 160 beats per minute. This routine will be undertaken five times a week, continuously for a span of 8 weeks.
  Interventions: Behavioral: Vigorous intermittent lifestyle physical activity

INTERVENTIONS:
Behavioral: Vigorous intermittent lifestyle physical activity — The specific exercise regimen involves performing rope jumping activities three times a day, with each session aimed at surpassing the exercise threshold (not conducted in a continuous manner), where the heart rate should exceed 160 beats per minute. This routine will be undertaken five times a week, continuously for a span of 8 weeks.

SUMMARY:
The goal of this clinicaltrial is to assess and compare isokinetic performance, surface electromyography, laboratory parameters, and cardiorespiratory function both before and after engaging in vigorous intermittent lifestyle physical activity(VILPA) within a healthy population.

The main question it aims to answer is:

[1] Does VILPA yield effective outcomes? Throughout the course of the trial, participants will engage in a simulated regimen of vigorous intermittent lifestyle physical activity for a duration of 8 weeks. The efficacy of the exercise protocol will be quantified and evaluated through the utilization of a wearable device.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Adults
* No exercise habits (more than 3 months)

Exclusion Criteria:

* Exercising ≥ 3 times per week;
* the presence of chronic diseases, such as hypertension, hyperglycemic states, etc;
* have conducted an exercise program in the past three months.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-05-12 (Actual); Primary Completion 2023-07-10 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Isokinetic strength testing | 30 minutes
  Isokinetic strength testing with the Isomed 2000
Surface electromyography | 15 minutes
  a standard surface electromyography system (MyoMove-EOW, NCC, China) was utilized. Surface electrodes were placed using the belly tendon method at 6 specified locations on both sides of the lower legs (anterior tibialis on both sides, gastrocnemius on both sides, and soleus on both sides). The electrode placement positions and operational procedures strictly adhered to the SENIAM guidelines (http://www.seniam.org). During the testing process, root mean square (RMS) and averaged electromyography (AEMG) values were collected to reflect the muscle force and motor unit recruitment of the selected muscle groups.

SECONDARY OUTCOMES:
Blood lipid | 5 minutes
  encompassing high-density lipoprotein cholesterol (HDL-C) and triglycerides, were assessed using the CardioChek device (Polymer Technology Systems, Inc., 7736 Zionsville Road, USA)

CONTACTS AND LOCATIONS:
Overall Officials: Lizhen Liao, Dr., Study Director — Department of Health, Guangdong Pharmaceutical University
Locations (1):
- Guangdong Pharmaceutical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No